CLINICAL TRIAL: NCT07406048
Title: A Real-World Study Evaluates the Clinical Characteristics and Effectiveness of COPD Patients Treated With the Triple Combination Beclometasone Diproprionate/Formoterol Fumarate/Glycopyrronium Bromide (BDP/FF/GB) in a Single Pressurised Metered Dose Inhaler (Trimbow® pMDI) in Brazil
Brief Title: Real-World Effectiveness of a Triple Combination BDP/FF/GB Extrafine in a Single Pressurised Metered Dose Inhaler in Brazilian COPD Patients
Acronym: RETRIBUTE
Status: Not yet recruiting | Type: Observational
Sponsor: Chiesi Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Other Study IDs: CLI-05993AA1-24
Record Dates: First submitted 2026-01-13; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; Real-world evidence; extra-fine particule; Trimbow; Fixed Triple Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trimbow: Adult patients with COPD treated with triple combination Beclometasone Diproprionate/Formoterol Fumarate/Glycopyrronium Bromide (BDP/FF/GB) as per local clinical practice
  Interventions: Drug: BDP/FF/GB (100ug/6ug/12.5ug)

INTERVENTIONS:
Drug: BDP/FF/GB (100ug/6ug/12.5ug) — Fixed combination of Inhaled Corticosteroid (ICS) / Long-acting β2-agonist (LABA) / long-acting muscarinic antagonist (LAMA) that contains Beclometasone dipropionate (BDP), Formoterol fumarate (FF) and Glycopyrronium bromide(GB)
  Other Names: Trimbow

SUMMARY:
This multicenter, retrospective-prospective, cohort study aims to evaluate the effectiveness and safety of Extra-fine Beclometasone Diproprionate/Formoterol Fumarate/Glycopyrronium Bromide (EF-BDP/FF/GB) therapy in adults with severe or very severe COPD in Brazil. Around 400 patients will be enrolled across approximately 15 sites. Eligible patients must have started treatment on the day of enrollment or up to three months before enrollment. Data will be collected both retrospectively and prospectively, with baseline information covering up to 12 months before treatment initiation. All assessments will occur during routine medical visits, with follow-up expected at approximately 3 ± 1 month and 6 months ± 2 months. The medication Trimbow® will not be provided as part of the study and must be prescribed and used according to the institution's standard clinical practice, regardless of participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients ≥ 40 years old at the time of BDP/FF/GB initiation
* Patients with documented diagnosis of severe or very severe COPD prior to BDP/FF/GB initiation
* Patients with CAT total score ≥ 10 at baseline (at the time of BDP/FF/GB initiation or within the 12 months before treatment initiation*) *If no CAT total score is available on BDP/FF/GB initiation date)
* Patients with at least ≥ 1 COPD exacerbation within the previous 12 months before enrollment.
* Patients who started treatment with BDP/FF/GB within 3-months before signing the Informed Consent Form (ICF), or on the date of the ICF signature according to Trimbow® Summary of Product Characteristics (SmPC)
* Patients who are willing and able to give their written consent to participate in the study

Exclusion Criteria:

- Patient known to be participating in any interventional study during the study period and in the 3 months prior to BDP/FF/GB initiation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brazilian patients aged ≥ 40 years old, diagnosed with severe and very severe COPD and with a CAT total score ≥ 10 at baseline, under treatment or who will initiate BDP/FF/GB treatment without previous use of single- inhaler triple therapy. Inclusion and exclusion criteria are listed above.
Sampling Method: Non-Probability Sample
Enrollment: 396 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the CAT (COPD assessment test) total score vs baseline at month 6 | Baseline and 6 months (±2 months)
  The test has a score of 0 (minimum) - 40 (maximum); a lower score means a better outcome, and a higher score means a worse outcome.

SECONDARY OUTCOMES:
Assessment of the CAT (COPD assessment test) total score vs baseline at month 3 | Baseline and 3 months (±1)
Change of Forced Expiratory Volume in one second assessed via spirometry | Baseline and 6 months (±2)
  Absolute value and percent of predicted normal of the following parameter: Forced Expiratory Volume in one second [FEV1 (L), mean ± SD (standard deviation)]; Percent predict FEV1 [FEV1 (% pred), mean ± SD]
Change of Forced Vital Capacity assessed via spirometry | Baseline and 6 months (±2)
  Absolute value of the following parameter: Forced Vital Capacity [FVC (L), mean ± SD]
Change of FEV1/FVC ratio assessed via spirometry | Baseline and 6 months (±2)
  Absolute value of the following parameter: Forced Expiratory Volume in one second / Forced Vital Capacity ratio: mean ± SD
Change of Forced Expiratory Flow at 25-75% of forced vital capacity via spirometry | Baseline and 6 months (±2)
  Absolute value of the following parameter: Forced Expiratory Flow at 25-75% of forced vital capacity [FEV25-75 (%), mean ± SD]
Safety Measure | 6 months (±2)
  * Overall summary of adverse drug reactions (ADRs) will be presented the number of subjects and percentage of subjects with any ADRs, including suspected ADRs and serious ADRs;
  * Overall summary of serious adverse events (SAE) will be presented the number of subjects and percentage of subjects with any SAE.
Descriptive statistics | Baseline and 6 months (±2)
  Patient profile - Descriptive statistics of :
  1. Demographic Data: Age; Sex; and State/region of residence.
  2. Clinical characteristics
     * Smoking history
     * COPD characteristics
     * Relevant medical history
     * COPD treatment
     * Concomitant medications
     * Vital signs

CONTACTS AND LOCATIONS:
Overall Officials: ROBERTO STIRBULOV, PhD, MD, Study Chair — Faculdade de Ciências Médicas da Santa Casa de São Paulo (FCMSCSP)

IPD SHARING:
Plan to Share IPD: No